CLINICAL TRIAL: NCT04949087
Title: Prospective, Double Blind, Randomized Control Trial Comparing the Efficacy of Intra-articular Injections for the Treatment of Primary Glenohumeral Osteoarthritis
Brief Title: Efficacy of Intra-articular Injections for the Treatment of Primary Glenohumeral Osteoarthritis(GHOA)
Acronym: GHOA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ORA 18060603
Record Dates: First submitted 2020-12-11; First posted 2021-07-02 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Arthritis Shoulder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-blinded, randomized
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Corticosteroid Injection Group (Experimental): 80mg Depo-Medrol and 8cc Lidocaine ultrasound-guided intra-articular injection
  Interventions: Procedure: Glenohumeral Injection
- Platelet-Rich Plasma Injection Group (Active Comparator): 15cc blood draw in Arthrex Autologous Conditioned Plasma (ACP) kit and processed per manufacturer instructions Ultrasound-guided intra-articular injection of isolated PRP
  Interventions: Procedure: Glenohumeral Injection

INTERVENTIONS:
Procedure: Glenohumeral Injection — Patients who enroll will be randomized into an injection group, and then will undergo the specified injection at one time point only.

SUMMARY:
The purpose of this study is to compare the efficacy of intra-articular corticosteroid injections versus platelet-rich plasma injections for non-operative treatment of primary glenohumeral osteoarthritis. The efficacy of intra-articular injections, outside of hyaluronic acid, for the treatment of glenohumeral OA is not known, yet these treatments are commonly used with hopes of providing patients with symptomatic relief that can hopefully delay or prevent the need for shoulder arthroplasty. This study will help elucidate the therapeutic benefit of corticosteroid and Platelet Rich Plasma (PRP) injections in this patient population.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥18y.o. of age
* Primary glenohumeral arthritis (bone on bone or near bone on bone) that has been previously diagnosed on radiographs and clinical evaluation.
* Baseline pain level of VAS >4

Exclusion Criteria:

* Secondary causes of arthritis (i.e. septic arthritis, rheumatoid arthritis, rotator cuff arthropathy, post-traumatic arthritis)
* Ipsilateral shoulder surgery within 1 year
* Any glenohumeral joint injection within 3 months
* Allergy to lidocaine
* Known pregnancy
* Workers compensation case regarding shoulder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-03-13 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale-Pain (VAS) | 12 weeks
  Validated patient-reported metric scale of pain: no pain (0-4 mm), mild pain(5-44 mm), moderate pain (45-74 mm), and severe pain (75-100 mm)

CONTACTS AND LOCATIONS:
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2020-07-30): https://cdn.clinicaltrials.gov/large-docs/87/NCT04949087/ICF_000.pdf